CLINICAL TRIAL: NCT00123812
Title: Frequency of Portal Images Required to Enhance Quality Assurance for Breast Cancer Patients Treated With Radiotherapy
Status: Withdrawn | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: BR-01-0056
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
Keywords: quality assurance; frequency of port films
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Currently in Canada, and at the Cross Cancer Institute, the treatment of many women with breast cancer involves radiotherapy (RT). There is a complex process which takes place in order to plan the radiation therapy before patients commence their treatment. In many circumstances the investigators use computerized technology to assist in planning their treatment. This allows more precision in delivering the treatment to the desired areas and avoiding areas of normal tissue.

Once the planning process is completed, the investigators then place marks with a marker pen on the skin of the patient to outline the area where the radiation will be delivered. The investigators confirm that the correct area is being treated with an x-ray taken on the treatment unit while the patient is in the treatment position. This is called a port film or verification film. The investigators then compare this to what they set up with the computerized data. If all the information matches, the patient is then treated for the full course of radiation, with the assumption that all treatments are given in the correct position. No further routine checking is done.

The standard at some radiotherapy centers is that the patient treatment position is verified weekly by a portal film. At the Cross Cancer Institute the investigators normally only do it once at the beginning of treatment.

No information is available to confirm the necessity of doing more frequent verification films, but in view of the very complex nature of the investigators' treatment delivery, it may be necessary to confirm the accuracy of their treatment more often.

Over the course of a 4-5 week treatment the investigators know that some patients may lose weight, some become more relaxed after a few days, and some have trouble with the movement in their shoulders; all of these factors influence the positioning of the patient. Measurements taken on the treatment unit often change during the course of a patient's treatment, but no further verification is performed to ensure that the treated area is still what was initially intended. It is important from a quality assurance standpoint to see if more frequent checking of the radiation treatment set-up is indicated.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

To determine if the verification film (port film) taken and accepted as correct at the beginning of a course of radiotherapy is adequate to ensure accurate position of treatment delivery for a 4-5 week course of radiotherapy in breast cancer patients.

Secondary:

* To assess the feasibility of doing on line portal imaging for breast cancer radiotherapy treatment.
* To possibly identify a patient population that should be verified daily with on line portal imaging.

DISCUSSION:

Quality assurance is a very important aspect of radiotherapy delivery. There are many facets of quality assurance but a basic concept is to ensure the radiation is delivered to the correct target area. At the start of a course of radiotherapy treatment the standard at the Cross Cancer Institute is to confirm the correct area is being treated. This is done by taking an x-ray on the treatment unit with the patient in the treatment position (portal image or verification film). This portal image is examined by the treating oncologist and compared to the simulation film or a digitally reconstructed radiograph that was generated when the patient was simulated (set up) for radiotherapy treatment. Some alterations may be suggested by the oncologist but once a portal film is deemed to reflect the original set-up - no more routine verifications are performed. It is assumed that the treatment set-up will be accurate for the remainder or the treatments.

Numerous changes may occur when a patient undergoes a 4-5 week course of RT. The patient may relax after a few treatments, a patient can lose weight, surgical changes can settle, all altering the original set up.

There are no data to determine how often a set up should be verified. Ideally it should be checked daily prior to each treatment initiation. This can be done with on line portal imaging however resources currently do not allow on line portal imaging for every patient. By evaluating the impact of weekly portal images the investigators may be able to identify a population of patients that would benefit from more frequent portal images or patients who would benefit from daily on line portal images, allowing for appropriate resource allocation.

Currently in Canada, and at the Cross Cancer Institute, the treatment of many women with breast cancer involves radiotherapy. There is a complex process which takes place in order to plan the radiation therapy before patients commence their treatment. In many circumstances the investigators use computerized technology to assist in planning their treatment. This allows more precision in delivering the treatment to the desired areas and avoiding areas of normal tissue.

Once the planning process is completed, the investigators then place marks with a marker pen on the skin of the patient to outline the area where the radiation will be delivered. The investigators confirm that the correct area is being treated with an x-ray taken on the treatment unit while in the treatment position. This is called a port film or verification film. The investigators then compare this to what they set up with the computerized data. If all the information matches, the patient is then treated for the full course of radiation, with the assumption that all treatments are given in the correct position. No further checking is done.

The standard at some radiotherapy centers is that the patient treatment position is verified weekly by a portal film. At the Cross Cancer Institute the investigators only do it once at the beginning of treatment.

No information is available to confirm the necessity of doing more frequent verification films, but in view of the very complex nature of the investigators' treatment delivery, it may be necessary to confirm the accuracy of their treatment more often.

Over the course of a 4-5 week treatment the investigators know that some patients may lose weight, some become more relaxed after a few days, and some have trouble with the range of movement in their shoulders; all of these factors influence the positioning of the patient. Measurements taken on the treatment unit often change during the course of a patients treatment, but no further verification is performed to ensure that the treated area is still what was initially intended.

STUDY DESIGN:

This is a single institute pilot project.

PATIENT CRITERIA/SAMPLE SIZE:

Any breast cancer patients receiving a course of radiotherapy to treat the breast, chest wall and/or regional lymph nodes.

One-hundred consecutive consenting patients will be analyzed prospectively. Patients will be stratified as per treatment area: breast only, breast plus regional nodes, chest wall only and chest wall plus regional nodes. The treatment technique will also be evaluated.

METHODOLOGY:

Patients eligible and consenting will be sequentially selected to undergo the standard radiotherapy planning process and initial verification films. In addition to the standard initial verification films, all patients will have additional verification films taken weekly. These will be reviewed by the treating radiation oncologist and a data form will be completed. The treatment record will also be examined and any changes noted by the therapists during the course of radiotherapy will be recorded.

No additional amount of radiation is given to the patient. The amount of radiation required to take the verification films is subtracted from the amount of radiation delivered at the time of treatment.

The data will be compiled and compared to establish any relationship between target volume (breast only, breast plus regional nodes, chest wall only and chest wall plus regional nodes) or technique used to the acceptability rate and accuracy of the verification films.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-03; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Susan Chafe, MD, Principal Investigator — Cross Cancer Institute